CLINICAL TRIAL: NCT03855943
Title: Personalized Computerized Inhibitory Control Training for OCD
Brief Title: Evaluating the Effects of a Computerized Training Program Coupled With Cognitive Behavioral Therapy (CBT) for OCD.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Noa Tauber, Research Assistant, Hebrew University of Jerusalem
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISF 1341/18
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT + Personalized Computer Program (Experimental): Cognitive Behavioral Therapy (CBT), consisting of Exposure and Ritual Prevention Therapy and training with a personalized computerized inhibitory training program
  Interventions: Behavioral: Personalized Computer Program; Behavioral: CBT

INTERVENTIONS:
Behavioral: Personalized Computer Program — Training with a personalized computerized inhibitory training program
Behavioral: CBT — Cognitive Behavioral Therapy (CBT), consisting of Exposure and Ritual Prevention Therapy

SUMMARY:
This study will evaluate the effects of a computerized training program coupled with cognitive behavioral therapy (CBT) for OCD.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of a computerized training program (called Personalized Computerized Inhibitory Training, or PCIT) coupled with cognitive behavioral therapies (CBT) consisting of Exposures and Response Prevention in treating obsessive compulsive disorder (OCD) in patients who previously underwent CBT, but still have residual symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of OCD (assessed by SCID).
* Clinically significant OCD symptoms (Y-BOCS score of at least 14).
* Allowed to be on medications if they have been on a stable dose for at least 12 weeks prior to the study and will remain on a stable dose during this study.
* Have access to a computer or laptop.

Exclusion Criteria:

* Individuals with the following disorders will excluded: bipolar, psychosis, current major depressive disorder (assessed by SCID).
* Patients with head injury and loss of consciousness of more than five minutes or a neurological condition affecting the central nervous system.
* Patients taking a psychiatric medication will be asked to maintain a stable dose for 6 weeks prior to study entry.
* Patients with a history of more than 8 hours of therapist-assisted ERP for OCD in the past 6 months,
* Vision or hearing loss (although individuals with vision corrected by glasses or contacts will not be excluded).
* Active suicidality warranting immediate clinical care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Obsessive-compulsive symptoms measured after 3 weeks of treatment | 3 weeks
  Measured by Yale-Brown Obsessive Compulsive Scale (YBOCS), considered the gold standard assessment tool.
  Y-BOCS comprises a Symptom Checklist and Severity Scale to consecutively rate obsessions and compulsions. The Checklist includes 54 common obsessions and compulsive behaviors, which are grouped according to thematic content. Symptoms that are endorsed over the past week are then globally rated by the clinician using a five-point scale ranging from 0 (none) to 4 (extreme) across five dimensions: (1) time/frequency, (2) interference, (3) distress, (4) resistance, and (5) degree of control. Obsessive and compulsive symptom severity are rated separately (scores range from 0 to 25) with these scores summed to create a total OCD severity score (range, 0-50).
  Symptom severity scores: mild symptoms (0-13), moderate symptoms (14-25), moderate-severe symptoms (26-34), and severe symptoms (35-40).26

CONTACTS AND LOCATIONS:
Overall Officials: Noa Tauber, MA, Principal Investigator — Hebrew University of Jerusalem
Locations (1):
- Hebrew University of Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No